CLINICAL TRIAL: NCT05569590
Title: Effiacacy of Desensitizing Agent,After an In-office Vital Tooth Bleaching. A Randomized Double Blind Clinical Trial Trial.
Brief Title: Efficacy of Desensitizing Agent,Propolis After an In-office Vital Tooth Bleaching.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Fatima Soomro, Efficacy of desensitizing agent Propolis,after an in-office vital tooth bleaching., Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FSoomro
Record Dates: First submitted 2022-09-28; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Post Operative Pain
Keywords: Tooth discoloration, vital tooth bleaching, dentine hypersensitivity, desensitizing agent, Propolis; Vital tooth bleaching
MeSH Terms: conditions — Pain, Postoperative; Tooth Discoloration; Dentin Sensitivity | interventions — Propolis

STUDY DESIGN:
Intervention Model Description: Subjects are randomly placed into one of the groups: Control, Propolis and Propolis mixed with bleaching agent. In Propolis group Propolis paste will be applied for 10 minutes. Post operative sensitivity will be assessed for 7 days by using visual analogue and Shiff's scale.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (participant, Outcome assessor) It is double blinded study in which participant will be blinded. the assessor who will assess the post operative sensitivity of the participant will also be blinded regarding the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): One visit three application of bleaching agent (hydrogen peroxide 35%) will be performed and desensitizing agent (fluoride varnish) will be applied for 10 minutes after bleaching.
  Interventions: Drug: hydrogen peroxide 35%; Other: fluoride varnish
- Propolis (Experimental): One sitting vital tooth bleaching procedure will be performed. Three application each of 15 minutes of bleaching agent (hydrogen peroxide 35%) will be applied and desensitizing agent propolis in paste form will be applied for 10 minutes.
  Interventions: Drug: Propolis; Drug: hydrogen peroxide 35%
- Propolis mixed with bleaching agent (Experimental): One visit vital tooth bleaching procedure will be performed. three application each of 15 minutes of Propolis mixed with bleaching agent (hydrogen peroxide 35%) will be applied.
  Interventions: Drug: Propolis; Drug: hydrogen peroxide 35%

INTERVENTIONS:
Drug: Propolis — Vital tooth bleaching will be performed and Propolis as a desensitizing agent will be applied after bleaching to reduce dentine hypersensitivity.
  Arms: Propolis; Propolis mixed with bleaching agent
Drug: hydrogen peroxide 35% — hydrogen peroxide 35%
Other: fluoride varnish — fluoride varnish
  Arms: Control

SUMMARY:
This study was conducted to evaluate the efficacy of desensitizing agent Propolis, after an in -office vital tooth bleaching and to compare its desensitizing effect to traditionally used desensitizing agent fluoride varnish.

Methods: Considering the inclusion and exclusion criteria 90 patients will be selected at the OPD of Dow University of Health Sciences Ojha campus with mild to moderate discoloration and randomly divided in to three groups group A control group (fluoride varnish) group B Propolis and group C Propolis mixed with bleaching agent. After performing the bleaching procedure respective desensitizing agent was applied to each group for 10 minutes. Visual analogue scale and Schiff's scale were used to assess the sensitivity after completion of treatment. Subjective non stimulated assessment of sensitivity was done by using the visual analogue scale from day 1 till day 7 on given Performa and Objective stimulated assessment of sensitivity was done at the dental office on day 1 right after the procedure and at day 7 on follow-up after one week.

Kruskal-Wallis test was applied to check median pain score and sensitivity difference between and among the groups. Mann-Whitney U test was applied to check further pairwise comparison between the groups.

DETAILED DESCRIPTION:
Dental aesthetic is one of the great importance to the patients, various causes of tooth discoloration which usually encountered are dental fluorosis, aging, staining, smoking, medication use, etc. Different treatment options are available to treat discoloration depends on the individual case. Dental bleaching is one of the most conservative, noninvasive, low cost effective treatment modality to treat discoloration. In vital tooth bleaching dentists use 35 to 38 % hydrogen peroxide which have the deleterious effects on tooth structures. The main problem which is usually experienced by the patients with the vital tooth bleaching is dentine hypersensitivity. Methods: Considering the inclusion and exclusion criteria 90 patients will be selected at the OPD of Dow University of Health Sciences Ojha campus with mild to moderate discoloration and randomly divided in to three groups group A control group (fluoride varnish) group B Propolis and group C Propolis mixed with bleaching agent. After performing the bleaching procedure respective desensitizing agent was applied to each group for 10 minutes. Visual analogue scale and Schiff's scale were used to assess the sensitivity after completion of treatment. Subjective non stimulated assessment of sensitivity was done by using the visual analogue scale from day 1 till day 7 on given Performa and Objective stimulated assessment of sensitivity was done at the dental office on day 1 right after the procedure and at day 7 on follow-up after one week.

Statistical analysis was carried out by using the software SPSS IBM version 26.Median and inter quartile range (IQR) were reported to describe continuous variables (pain and sensitivity score) Normality of continuous variable (VAS pain score and sensitivity score) was checked by using the Shapiro-wilk test and Kruskal-Wallis test was applied to check median pain score and sensitivity difference between the groups. Mann-Whitney U test was applied to check further pairwise comparison between the groups. Chi-squire test was applied and cross tabulation done to see the association between all groups and visual analog scale. P-values of less than or equal to ≤ 0.05 were used to determine the significance of all test results.

ELIGIBILITY:
Inclusion Criteria:

* • Presence of all anterior teeth with mild to moderate discoloration

  * Patient's age must be 18 to 30 years
  * Absence of pre-operative pain or sensitivity
  * Patients having no history of smoking
  * Patients with no cervical lesions and exposed roots
  * Good oral hygiene using simplified oral hygiene index
  * NO or minimum dental hypersensitivity to heat and cold before bleaching.

Exclusion Criteria:• Patients with any kind of restoration, calculus or heavy stain on study site

* Candidates with severe discoloration
* Gross pathology with in oral cavity
* The Presence of heavy stains or calculus on study sites.
* Patients using any analgesics
* Patients having the use of desensitizing agent in any form.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Assessment of efficacy of desensitizing agent Propolis after an in office vital tooth bleaching | Post operative sensitivity was assessed for 7 days after treatment. Visual analogue scale was used to assess the pain (sensitivity).
  Visual analogue scale (VAS) was used to assess the postoperative dentine hypersensitivity after procedure. Performa was provided to the patients which include VAS. the scale is usually a straight line 10 cm line which clearly defined boundries 0= no pain,1-3=mild pain,4-6 moderate pain and 7-10 severe pain.patients marked the no according to their pain ( sensitivity) level.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Soomro, MDS, Principal Investigator — DUHS
Locations (1):
- Fatima Soomro, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No